CLINICAL TRIAL: NCT04629105
Title: A Phase 1 Double-blinded, Randomized, Placebo-controlled Study for COVID-19 and Influenza Virus-Elicited Acute Respiratory Distress Syndrome (ARDS) Using Lomecel-B
Brief Title: Regenerative Medicine for COVID-19 and Flu-Elicited ARDS Using Lomecel-B (RECOVER)
Acronym: RECOVER
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Longeveron Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00-006
Record Dates: First submitted 2020-09-29; First posted 2020-11-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: ARDS, Human; Covid19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, placebo-controlled study with 2 cohorts.
  Cohort 1: Subjects with ARDS and acutely infected with SARS-CoV-2. Arm 1: 25 subjects treated with up to 3 doses of 100 million LMSCs. Arm 2: 10 subjects treated with up to 3 doses of Placebo.
  Cohort 2: Subjects with ARDS and acutely infected with influenza virus. Arm 3: 25 subjects treated with up to 3 doses of 100 million LMSCs. Arm 4: 10 subjects treated with up to 3 doses of Placebo.
  Each subject will be intravenously infused with 100 million LMSCs or placebo on Day 0. If no treatment-related AEs are seen after the infusion, a second infusion will be given on Day 3. If no treatment-related AEs are seen after the second infusion, a third infusion will be given Day 6.
  Follow-up visits will be conducted: daily until hospital discharge; at Week 4 after treatment (with LMSCs or placebo) for patients already discharged; and at Month 6 after treatment (with LMSCs or placebo).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (SARS-CoV-2): Arm 1 (LMSCs) (Active Comparator): Cohort 1: Subjects with ARDS and acutely infected with SARS-CoV-2. Arm 1: 25 subjects treated with up to 3 doses of 100 million LMSCs.
  Interventions: Biological: Longeveron Mesenchymal Stem Cells (LMSCs)
- Cohort (SARS-CoV-2): Arm 2 (Placebo) (Placebo Comparator): Cohort 1: Subjects with ARDS and acutely infected with SARS-CoV-2. Arm 2: 10 subjects treated with up to 3 doses of Placebo.
  Interventions: Other: Placebo
- Cohort 2 (Flu): Arm 3 (LMSCs) (Active Comparator): Cohort 2: Subjects with ARDS and acutely infected with influenza virus. Arm 3: 25 subjects treated with up to 3 doses of 100 million LMSCs.
  Interventions: Biological: Longeveron Mesenchymal Stem Cells (LMSCs)
- Cohort 2 (Flu): Arm 4 (Placebo) (Placebo Comparator): Cohort 2: Subjects with ARDS and acutely infected with influenza virus. Arm 4: 10 subjects treated with up to 3 doses of Placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Longeveron Mesenchymal Stem Cells (LMSCs) — Longeveron Mesenchymal Stem Cells (LMSCs)
  Arms: Cohort 1 (SARS-CoV-2): Arm 1 (LMSCs); Cohort 2 (Flu): Arm 3 (LMSCs)
Other: Placebo — Placebo
  Arms: Cohort (SARS-CoV-2): Arm 2 (Placebo); Cohort 2 (Flu): Arm 4 (Placebo)

SUMMARY:
A Phase I, double- blinded, randomized, placebo- controlled study to test the safety of Lomecel-B in Adults suffering from mild to severe acute respiratory distress syndrome (ARDS) due to COVID-19 resultant from 2019-nCoV coronavirus infection, or resultant from influenza virus infection.

DETAILED DESCRIPTION:
Double-blinded, randomized, placebo-controlled study with 2 cohorts.

Cohort 1: Subjects with ARDS and acutely infected with SARS-CoV-2. Arm 1: 25 subjects treated with up to 3 doses of 100 million Lomecel-B Arm 2: 10 subjects treated with up to 3 doses of Placebo.

Cohort 2: Subjects with ARDS and acutely infected with influenza virus. Arm 3: 25 subjects treated with up to 3 doses of 100 million Lomecel-B Arm 4: 10 subjects treated with up to 3 doses of Placebo.

Each subject will be intravenously infused with 100 million Lomecel-B (formerly LMSCs) or placebo on Day 0. If no treatment-related AEs are seen after the infusion, a second infusion will be given on Day 3. If no treatment-related AEs are seen after the second infusion, a third infusion will be given Day 6.

Follow-up visits will be conducted: daily until hospital discharge; at Week 4 after treatment (with LMSCs or placebo) for patients already discharged; and at Month 6 after treatment (with LMSCs or placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female or any race or ethnicity.
2. At least 18 years of age.
3. Provide written informed consent. For subjects who are incapable of providing informed consent, written informed consent can be provided on behalf of the subject by a legally authorized representative (LAR).
4. Diagnosis of mild to severe ARDS per the Berlin Definition of ARDS. More specifically, the following 3 conditions must be present.

   1. A need for positive pressure ventilation by an endotracheal or tracheal tube with a PaO2/FiO2 ratio < 200 with at least 8 cm H2O positive end-expiratory airway pressure (PEEP). A patient may be included if the PaO2/FiO2 ratio < 200 with < 8 cm H2O PEEP if there is a contraindication to increased PEEP (evidence of barotrauma).
   2. Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph.
   3. No clinical evidence of left atrial hypertension for bilateral pulmonary infiltrates.
5. Confirmed diagnosis of infection with coronavirus or influenza virus.
6. Willing to perform all assessments required for the study.
7. Must agree to the collection of all blood samples per protocol.
8. Must agree to have samples stored and used for secondary research.

Exclusion Criteria:

1. Patient receiving Extracorporeal Membrane Oxygenation (ECMO).
2. History of malignancy within previous 2.5 years, except for curatively-treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ, or cervical carcinoma.
3. Prior positive test for any of the following without demonstration of resolution.

   i. Hepatitis B virus (HBV) surface antigen (HBsAg). ii. Viremic hepatitis C virus (HCV). iii. Human immunodeficiency virus-1 or -2 (HIV1 or 2 HIV2). iv. Human T-cell leukemia virus-I or -II (HTLV-I or HTLV-II). v. Syphilis.
4. Female who is pregnant, nursing, or of childbearing potential while not practicing effective contraception.
5. Known hypersensitivity to dimethyl sulfoxide (DMSO).
6. Be an organ transplant recipient, other than for corneal, bone, skin, ligament, or tendon transplant.
7. Actively listing (or expected listing) for transplant of any organ, other than for corneal, bone, skin, ligament, or tendon transplant.
8. Continuous use of any medication at immunosuppressive dosing for greater than 14 consecutive days over the past 3 months.
9. Currently participating in an investigational therapeutic or device trial, or have participated in an investigational therapeutic or device trial within the previous 30 days, or participate in any other clinical trial for the duration of the time that the subject actively participates in this trial. However, use of hydroxychloroquine, remdesivir, lopinavir/ritonavir and ivermectin are allowed as well as convalescent plasma.. Exceptions for other experimental interventions related to treating the patient's acute illness may be made with prior approval of Longeveron.
10. Any serious comorbid illness or any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study, or that may compromise the validity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Serious Adverse Events | Within 4 weeks after treatment
  Incidence of treatment-emergent serious adverse events (TE-SAEs) within 4 weeks after treatment, defined as one or more of the following untoward medical occurrences happening within the first 4 weeks after treatment.
  i. Life-threatening event (e.g., stroke or non-fatal pulmonary embolism). ii. Event requiring inpatient hospitalization or prolongation of existing hospitalization (e.g., for worsening dyspnea).
  iii. Event resulting in persistent or significant disability/incapacity. iv. Event resulting in death. v. Event leading to other clinically significant untoward laboratory test result(s) or medical condition(s), as determined by the Investigator.
Number of Participants with Abnormal Clinical Significant Laboratory Values in Hematology. | Baseline to 6 Months
  Number of Participants with Abnormal Clinical Significant Lab Values in the Hematology testing will be assessed at Baseline and 6 Months.
Number of Participants with Changes in Echocardiography Overall Assessment | Baseline to 6 Months
  Overall Assessment Normal vs Abnormal will be collected at Baseline and 6 months, this change in overall assessment will be the outcome in numbers of particants with a change.
Number of Participants with Changes to overall assessment of Electrocardiogram | Baseline to 6 Months
  Number of Participants with changes to Overall Assessment Normal vs Abnormal will be collected at Baseline and 6 Months
Time to recovery of Sp02 | Baseline to 6 Months
  Time to recovery of Sp02 to 90% or higher on room air (or the oxygen concentration the patient had before acute illness) after 10 minutes of spontaneous breathing.
Number of Participants with Abnormal Clinical Significant Lab Values in the Blood Chemistry testing. | Baseline to 6 months
  Number of Participants with Abnormal Clinical Significant Lab Values in Blood Chemistry testing will be assessed at Baseline and 6 Months.
Number of Participants with Abnormal Clinical Significant Lab Values in the Coagulation. | Baseline to 6 months
  Number of Participants with Abnormal Clinical Significant Lab Values in the Coagulation testing will be assessed at Baseline and 6 Months.
Number of Participants with Abnormal Clinical Significant Lab Values in the Urinalysis | Baseline to 6 months
  Number of Participants with Abnormal Clinical Significant Lab Values in the Hematology testing will be assessed at Baseline and 6 Months.

SECONDARY OUTCOMES:
Immunity | Baseline to 6 Months
  Geometric mean titer
Change in Imaging via X-ray | Baseline to 6 Months
  Change in overall assessment via Lung imaging via chest X-ray will be assessed and compared between baseline and 6 months
Change in Imaging via Computerized Tomography | Baseline to 6 Months
  Change in overall assessment via Lung imaging via computerized tomography will be assessed and compared between baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Miami VA Healthcare System, Miami, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina